CLINICAL TRIAL: NCT01392547
Title: Efficacy and Safety of NNC 0078-0000-0007 in Treatment of Acute Bleeding Episodes in Patients With Congenital Haemophilia and Inhibitors
Brief Title: Efficacy and Safety of NNC 0078-0000-0007 in Patients With Congenital Haemophilia and Inhibitors
Acronym: adept™2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1731-3562; 2010-023803-92 (EudraCT Number); U1111-1118-2228 (Other: WHO); JapicCTI-111595 (Registry Identifier: JAPIC)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2015-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — vatreptacog alfa; Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFVIIa (Experimental)
  Interventions: Drug: eptacog alfa (activated)
- vatreptocog alfa (Experimental)
  Interventions: Drug: vatreptacog alfa (activated)

INTERVENTIONS:
Drug: vatreptacog alfa (activated) — 1-3 doses per bleeding episode
  Arms: vatreptocog alfa
Drug: eptacog alfa (activated) — 1-3 doses per bleeding episode
  Arms: rFVIIa

SUMMARY:
This trial is conducted globally. The purpose of this trial is to confirm the efficacy and safety of NNC 0078-0000-0007 in patients with congenital haemophilia and inhibitors.

DETAILED DESCRIPTION:
Scheduled dose visit in a non-bleeding state. Single dose of NNC 0078-0000-0007 (vatreptocog alfa (activated)) every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male patient with clinical diagnosis of congenital haemophilia A or B and inhibitors to coagulation factors VIII or IX
* Minimum of five bleeds requiring haemostatic drug treatment within the previous 12 months at trial entry

Exclusion Criteria:

* Previous participation in this trial defined as withdrawal after administration of trial product
* Patient has received an investigational medicinal product within 30 days prior to this trial
* Congenital or acquired coagulation disorders other than haemophilia A or B
* Any clinical signs or known history of arterial thrombotic events or of deep venous thrombosis or pulmonary embolism (as defined by available medical records)
* Platelet count of less than 50,000 platelets/mcL (at the screening visit)
* ALAT (alanine-transaminase) of more than 3 times the upper normal limit (according to laboratory reference ranges)
* Factor VIII/IX Immune Tolerance Induction regimen planned to occur during the trial
* Ongoing bleeding prophylaxis regimens or planned bleeding prophylaxis to occur during the trial
* HIV (Human Immunodeficiency Virus) positive with current CD4+ count of less than 200/mcL (defined by medical records)

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (31):
- United States (13):
  - Novo Nordisk Clinical Trial Call Center, Tucson, Arizona
  - Novo Nordisk Clinical Trial Call Center, Los Angeles, California
  - Novo Nordisk Clinical Trial Call Center, Orange, California
  - Novo Nordisk Clinical Trial Call Center, Aurora, Colorado
  - Novo Nordisk Clinical Trial Call Center, Tampa, Florida
  - Novo Nordisk Clinical Trial Call Center, Atlanta, Georgia
  - Novo Nordisk Clinical Trial Call Center, Augusta, Georgia
  - Novo Nordisk Clinical Trial Call Center, Iowa City, Iowa
  - Novo Nordisk Clinical Trial Call Center, Boston, Massachusetts
  - Novo Nordisk Clinical Trial Call Center, Detroit, Michigan
  - Novo Nordisk Clinical Trial Call Center, Brooklyn, New York
  - Novo Nordisk Clinical Trial Call Center, Portland, Oregon
  - Novo Nordisk Clinical Trial Call Center, Richmond, Virginia
- Linz, Austria
- Campinas, São Paulo, Brazil
- Zagreb, Croatia
- Athens, Greece
- Budapest, Hungary
- Milan, Italy
- Shinjuku-ku, Tokyo, Japan
- Kuala Lumpur, Malaysia
- Warsaw, Poland
- Novo Nordisk Clinical Trial Call Center, San Juan, Puerto Rico
- Timișoara, Timiș County, Romania
- Saint Petersburg, Russia
- Novi Sad, Serbia
- Parktown, Johannesburg, Gauteng, South Africa
- Changhua, Taiwan
- Bangkok, Thailand
- Bornova-IZMIR, Turkey (Türkiye)
- Oxford, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients treated with vatreptacog alfa were recruited from a total of 46 sites globally in 18 countries, including Austria, Brazil, Croatia, Greece, Hungary, Italy, Japan, Malaysia, Poland, Romania, Russia, Serbia, South Africa, Taiwan, Thailand, Turkey, United Kingdom and United States of America.
Groups:
- Vatreptacog Alfa and rFVIIa (All Subjects): Subjects participating in the trial were randomised to receive vatreptacog alfa and rFVIIa in a cross-over manner. Subjects participating in the trial had bleeding episodes randomised to treatment with either vatraptacog alfa or rFVIIa in an independent manner for each bleeding episodes. Of the 72 subjects, 3 subjects did not have any bleeds.
Period: Overall Study
Arm/Group | Vatreptacog Alfa and rFVIIa (All Subjects)
Started | 72 (567 bleeds by 69 subjects, 340 were treated with vatreptacog alfa and 227 with rFVIIa)
Completed | 64
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Non-compliance | 2
Not completed — Withdrawal criteria | 3
Not completed — Unclassified | 1

BASELINE CHARACTERISTICS:
Groups:
- Vatrepcacog Alfa and rFVIIa: Subjects participating in the trial were randomised to receive vatreptacog alfa and rFVIIa in a cross-over manner.
Arm/Group | Vatrepcacog Alfa and rFVIIa
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.19 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Effective Bleeding Control Defined as no Additional Haemostatic Medication (Other Than Trial Product) Given
Time Frame: Within 12 hours of first trial product administration
Population: Patients with ≥1 efficacy data point. 567 bleeds in 69 patients were treated with vatreptacog/rFVIIa in random sequence. Bleeds excluded in case of identical consecutive treatments, use of both trial products, unknown dispensing unit number.
Measure: Number; unit: bleeding episodes
Groups:
- Vatreptacog Alfa 80 µg/kg: Vatreptacog alfa was administered intravenous bolus, 1-3 doses at 80 µg/kg body weight until haemostasis was achieved for a bleed
- rFVIIa 90 µg/kg: Recombinant factor VIIa (rFVIIa) was administered intravenous bolus, 1-3 doses 90 µg/kg body weight until haemostasis was achieved for a bleed
Arm/Group | Vatreptacog Alfa 80 µg/kg | rFVIIa 90 µg/kg
Number analyzed (Participants) | 67 | 57
bleeding episodes
  Additional haemostatic given | 22 | 16
  Additional haemostatic not given | 318 | 211

2. Secondary Outcome: Effective and Sustained Bleeding Control
Time Frame: Up to 48 hours after first trial product administration
Population: as for outcome 1
Measure: Number; unit: bleeding episodes
Arm/Group | Vatreptacog Alfa 80 µg/kg | rFVIIa 90 µg/kg
Number analyzed (Participants) | 67 | 57
bleeding episodes
  Additional haemostatic given | 53 | 51
  Additional haemostatic not given | 268 | 163

3. Secondary Outcome: Number of Doses of Trial Product Given for Each Acute Bleed
Time Frame: Up to 6 hours after first trial product administration
Population: as for outcome 1
Measure: Number; unit: bleeding episodes
Arm/Group | Vatreptacog Alfa 80 µg/kg | rFVIIa 90 µg/kg
Number analyzed (Participants) | 67 | 57
bleeding episodes
  1 dose | 51 | 23
  2 doses | 94 | 62
  3 doses | 195 | 142

4. Secondary Outcome: Number of Adverse Events
Description: Any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Adverse events were captured from the time of consent to 1 month (+14 days) after last administration of trial product.
Population: All patients exposed to at least one dose of trial product was included in the safety analysis set. Patients received scheduled doses with rFVIIa, and treatment (rVIIa and vatreptacog alfa) for each bleeding episode.
Measure: Number; unit: events
Arm/Group | Vatreptacog Alfa 80 µg/kg | rFVIIa 90 µg/kg
Number analyzed (Participants) | 72 | 57
events
  All adverse events | 55 | 11
  Mild adverse events | 33 | 5
  Moderate adverse events | 15 | 2
  Severe adverse events | 7 | 4

5. Secondary Outcome: Immunogenicity (Inhibitor Development)
Description: Immunogenicity was tested by formation of neutralising antibodies towards vatreptacog alfa and/or FVII. Radioimmunoassay using [125I]-labelled vatreptacog alfa or rFVIIa was used to screen plasma samples for development of anti-drug antibodies
Time Frame: Adverse events were captured from the time of consent to the end of trial visit 1 month (+14 days) after last administration of trial product.
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Vatreptacog Alfa 80 µg/kg | rFVIIa 90 µg/kg
Number analyzed (Participants) | 72 | 57
Subjects
  Positive for anti-vatreptacog alfa | 8 | 0
  Cross-reactive with rFVIIa | 4 | 0
  Positive for anti-rFVIIa | 0 | 1
  In vitro vatreptacog alfa-neutralising | 1 | 0
  In vitro FVII/rFVIIa-neutralising | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of consent to 1 month (+14 days) after last administration of trial product.
Description: All patients exposed to at least one dose of trial product was included in the safety analysis set.
Arm/Group | Vatreptacog Alfa 80 µg/kg | rFVIIa 90 µg/kg
Serious Adverse Events (participants affected / at risk) | 4/72 | 4/57
Other Adverse Events (participants affected / at risk) | 5/72 | 3/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatreptacog Alfa 80 µg/kg (N=72) | rFVIIa 90 µg/kg (N=57)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatreptacog Alfa 80 µg/kg (N=72) | rFVIIa 90 µg/kg (N=57)
Drug specific antibody present (Investigations) | 5 (8) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.